CLINICAL TRIAL: NCT03614104
Title: Awareness Development and Usage of mHealth Technology Among Hypertensive Patients in a Rural Community of Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Responsible Party: Principal Investigator, Yasmin Jahan, Principal Investigator, Hiroshima University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18H03111300
Record Dates: First submitted 2018-07-27; First posted 2018-08-03 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Hypertension
Keywords: Mobile health technology
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobile health technology (Active Comparator): Health education with mobile health technology
  Interventions: Behavioral: Mobile Health Technology (short message service)
- Without mobile health technology (Sham Comparator): Health education without mobile health technology
  Interventions: Behavioral: Mobile Health Technology (short message service)

INTERVENTIONS:
Behavioral: Mobile Health Technology (short message service) — Health education through mobile technology with Short Message Service (SMS)

SUMMARY:
To develop awareness, enhance knowledge, attitude and make behavioral changes by using health education and mHealth technology among hypertensive patients in a rural community of Bangladesh, A Randomized Controlled Trial will be conducted in a rural community around Kumudini Women's Medical College and Hospital, Mirzapur, Bangladesh, intervention period will be consecutive 5 months and 210 in each group (total 420). Face to face interviews will be conducted to develop awareness among hypertensive individuals as part of the provision of improved health care services. The face to face interview will take place at Kumudini Hospital or in the community. Face to face interviews will help to understand the individuals' perceptions, attitudes, and practices associated with compliance to treatment and behavior change. Additionally, the study will identify major barriers related to hypertension associated with healthcare-seeking behaviors. Subjects will be diagnosed cases of hypertension. The selection criteria would be: individuals aged 35 years and more, have at least 1-5 years of schooling, who are open and can exchange their views freely as well as who can be asked in-depth and probing questions. Moreover, specimens will be collected to examine for serum total cholesterol, random blood sugar, urinary salinity, and urinary protein. Physical measurements like height in meter, weight in kg, MUAC in millimeter, hip and waist ratio will be performed from the day of enrollment till the end of follow up. If the participant agrees to participate, they will be asked questions about their lifestyle, present health status, and socio-demographic characteristics. The interview will around 30 minutes of their time, measurement of nutritional status (height, weight, MUAC, hip circumference, and waist circumference), and specimen collection for laboratory tests (blood and urine) will take another 30 minutes. Initially, the follow-up visits will be twice a month then once a month up to 4 consecutive months. Interviews will be conducted in the Kumudini Women's Medical College and Hospital. The data will be securely stored in a locked room. Data will be processed and analyzed by using the statistical software packages SPSS for Windows version 21.0 and Epi Info version 6.0. Statistical significance will be defined as p<0.05.

DETAILED DESCRIPTION:
Introduction:

Hypertension is one of the foremost non-communicable diseases (NCDs)c in the world, which significantly contributes to the burden of cardiovascular diseases (CVDs), stroke, kidney failure, disability, and premature death. It is also recognized as a global public health problem and ranked third as a cause of disability-adjusted life-years (DALYs). According to the World Health Organization (WHO), about 17 million deaths occur worldwide due to CVDs, of which hypertension alone accounts for 9.4 million deaths and 80% of the CVD-related deaths occurred in the developing countries. The global prevalence of hypertension is projected to increase from 26% in 2000 to 29% by 2025, which will be approximately 29% of the world's population. Its prevalence is increasing in the low and middle-income countries (LMIC), especially Southeast Asia where individuals are having an increasing burden of hypertension including CVDs. According to WHO, hypertension has become a significant health concern in the Asian region, affecting more than 35% of the adult population. Bangladesh, a developing country in South Asia, has been experiencing an epidemiologic transition from communicable diseases to NCDs. In recent years, rapid urbanization, prolonged life expectancy, unhealthy diet, and lifestyle changes have led to an increase in the rate of CVD including hypertension in Bangladesh. In recent years, in Bangladesh, approximately 20% of adults and 40-65% of elderly people suffer from HTN. Most of the common reasons are sedentary lifestyle, changing food habit, smoking, and adulteration of food products, fruits, and vegetables. However, keeping in mind the changes in lifestyle and food habits among the young adults in Bangladesh, the possibilities of hypertension in young adults can't be ruled out among this age group. In this study, we aim to develop awareness, enrich knowledge and make behavioral modifications by health education and mHealth technology among hypertensive patients in a rural community of Bangladesh.

Objectives:

General objective:

1. To develop awareness and enhance knowledge, which will be measured by actual behavioral changes by using health education and mHealth technology among hypertensive patients in a rural community of Bangladesh.

   Specific objectives:
2. To evaluate the level of blood pressure changes
3. To measure health status by Euro-5D-5L QOL questionnaire (Mobility, self-care, usual activities, pain/discomfort, anxiety/depression)
4. To decrease dietary salt intake (Measured by food and urinary salinity test)
5. To measure blood glucose level (Random Blood Sugar), urinary protein and glucose test to measure complications.
6. To evaluate the feasibility of this intervention strategies and mHealth technology.

Hypothesis:

Here we hypothesize that hypertensive patients because of health education and mHealth technology applications (cell phone monitoring of BP and periodic behavioral change education - drug adherence) and follow-up will have decreased blood pressure (BP) relative to controls under medication but without any mHealth technology applications. Compared to controls, intervention patients at follow-up will report quality of life, behavioral change, dietary habit as well as their greater satisfaction with care.

Sample size calculation In this study we have considered two groups, intervention group (PI; health education with text messaging) and control group (PC; health education without text messaging). In each group a proportion of the participants will respond to the intervention; PI and PC. When the intention of the study is to show that the intervention group is superior than the usual formulation of null hypothesis (PI>PC).

In this study the investigators want to compare between two interventions (health education with or without text messaging). Investigators regard the compliance as PI>PC. We assume that, if the proportion of patients with compliance is at most 10% to 12% better in the health education with text messaging group.

Sample size was calculated with 2-tailed 5% significance level, power 80% with a confidence level of 95% (1-α) and to detect varying differences in the effectiveness of the two intervention groups. Assuming adherence rates differing between 10-12% with 90% in the study group and 78%, 79% and 80% respectively in the control group and with a presumption that 6% of the participants would be lost during follow-up. The sample size was calculated to range between 153-210 in each group. Thus, considering the largest size of the calculated sample sizes, the study finally had a sample size of 210 in each group.

Randomization:

A randomization schedule is being prepared following a permuted block randomization technique using a block size of four based on a computer-generated series of numbers. An experienced researcher (third party), who is not involved with the study generated the random allocation by sequence and distributed that in serially numbered sealed opaque envelopes which are being kept in locked file cabinets in a site away from trial's location. Thus, all CHWs and the principal investigator (PI) are kept blinded about the random allocation. A total of eight CHWs are being involved in participants' enrollment under the guidance of the PI. Sequential ID numbers of the potential participants are arranged by the PI immediately before enrolling in the field on a daily basis. Enrollment takes place during morning hours for consecutive 6 days (except Friday) in a week. CHWs open the envelope in front of the participants at their household when they agree to be enrolled in the study by giving written informed consent.

Enrollment of participants:

The study will be implemented at Kumudini Women's Medical College and Hospital immediately after getting IRB approval from Bangladesh Medical and Research Council (BMRC). Hypertensive patients living in rural Mirzapur will be mostly identified from Mirzapur Kumudini Hospital. Additionally, study participants will be selected from the community by the door to door visits. The diagnosis of hypertension will be based on the prescription and Kumudini hospital database records.

Study Activities and Data Collection Procedure:

Qualitative study

The present qualitative assessment will follow an exploratory study design. The study will particularly aim to comprehend the knowledge level in relation to hypertension in a rural community of Bangladesh. To achieve the study objectives, this study will adopt focus group discussion (FGD), in-depth-interviews (IDI), and key informant interviews (KII). These tools are omnipresent in qualitative study and provide subjective perceptions from community and individual perspectives.

Target population The inclusion criteria of these specific predefined participants for KII and IDI will be as follows: (i) male and female individuals aged ≥35 years, (ii) diagnosed recently or before as a hypertensive or non-hypertensive individual through review of hospital logs, and prescriptions (iii) physically and intellectually able to travel, attend and talk in interviews and actively participate in discussions, and (iv) who can be asked probing questions, can share their knowledge, perception, attitude towards hypertension and mHealth technology freely.

Qualitative study sample size:

Following number of participants will be interviewed:

Data collection tools Number of participants Key informant interview 6-8 (3-4 M & 3-4 F) In-depth interview 6-8 (3-4 M & 3-4 F) FGD with hypertensive male and female participants 60-80 (30/40 M & 30/40 F)

Data collection

The data will be collected through individual interviews (key informant interviews) and group interviews (focus group discussions).

1. Focus group discussion (FGD)

   FGD will be conducted in individuals with and without hypertension including both male and females at the community level to understand their perceptions, symptoms, knowledge, motivations, beliefs and attitude towards hypertension and mHealth technology and their practices related to healthcare at household and community level.
2. In-depth interview (IDI)

   The in-depth interviews will be conducted with 3-/4 people with hypertension and 3-/4 people without hypertension both male and female who are individuals of either sex from local community to understand their perceptions, knowledge about symptoms of hypertension, motivations, beliefs and attitude towards hypertension and mHealth technology and their health care seeking practices and compliances towards drugs and instructions.
3. Key informant interview (KII)

In relation to the study objectives, the study will conduct key informant interviews to develop an insight of individuals regarding the symptoms, causes and consequences of hypertension, the importance of lifestyle modification and regular check-ups in controlling hypertension or barriers and challenges that keep them away from regular checkups and medication adherence. Moreover, the systems that affect mobile health related health care services at the local level, potential barriers and challenges, and issues that may need further attention will be identified.

Data Management and Analysis

Data from field will follow a step-by-step data management procedure:

1. Data labelling (naming the recorded and transcribed files)
2. Transcription (both in Bangla and English)
3. Data cleaning (recover missing data)
4. Data compilation with field notes (check the accuracy and brevity)
5. Data storage (both soft and hard copy in a safe and secure place with restricted access)

Data Analysis After having a good sense of field data, the research team will initiate a thematic/content analysis based on available data. Both inductive (bottom-up: emerging from field data) and deductive (top-down: theory driven) approach of coding and themes (/sub-themes) selection will be taken into consideration. However, it is important to note that data analysis in a qualitative study is consistent process rather than step-by-step.

Data coding At first, transcripts will be reviewed carefully and re-read for producing a code book. Reading and coding will initiate while data are being collected.

Data presentation The data display and reduction process will be conducted once all data have been collected. Even during data display and reduction, the investigators will loop back through earlier steps to refine codes, re-read texts and revise some aspects of analysis. After reading, re-coding and coding the text, the main themes will be formalized.

Enrollment of participants for RCT:

Immediately before the implementation of the research, a structured questionnaire will be developed based on past experience in rural Bangladesh and elsewhere, which will be discussed thoroughly with field staff members and extensive field-testing will be done for necessary modifications of the questionnaire. Using a standardized pre-tested questionnaire, the socio-economic status and demography ( age, sex, religion, financial dependency, educational qualification, occupation, monthly family income and expense, type of house, type of family, marital status, living arrangements and so on) health status, health care seeking behavior, food consumption practices, life styles such as tobacco consumption, level of physical activity and other relevant information will be obtained. Moreover, blood and urine specimens will be collected and laboratory tests like serum total cholesterol, random blood sugar, urinary salinity, and urinary protein, glucose will be performed. Measurements of nutritional indices such as height, weight, MUAC, hip circumference, and waist circumference will be carried out from the enrollment day till end of follow up. Follow up and physical examination will take place at Kumudini Hospital or in the nearest Health and Family Welfare Center. In this study, we will use a portable health clinic device which is recommended by Grameen health program and by using this device we can save our time, as this device has all the test and measurement facilities which we will do in our study. Six follow up visits will be undertaken during the study period. Initially follow up visits will be twice a month then once a month up to 4 consecutive months.

Moreover, staff members will be trained on use of all hardware. Usability evaluation of the staff members will be performed to document (a) user performance and understand common errors that are made by them while using the devices, (b) understand user perceptions and their suggestions in better usage of the devices. Similar usability evaluation of the 10-15 hypertensive individuals will be conducted. The evaluation will be conducted in a quiet environment with no distractions. Five qualitative questions will be asked to understand the practical benefits and drawbacks of the devices. SMS messages will be developed in native language by the members of the research team representing different professional background; these messages will be sent to 10-15 people (randomly) for their comprehension and acceptability as part of field-testing. The wired intervention individuals will receive short messaging service (SMS) and they will have liberty to participate additionally in two-way communication system (between wired individuals and research team members). After receiving feedback, messages will be finalized. The SMS will provide simple health education and BP measurement reminders to encourage adherence to medical advice. Research team members will send a text message to a wired person having registered cell phone number throughout the study period. SMS (First month: 3 SMS per week, and then third month to five months: 1 SMS per week).

All the enrolled patients will receive health education booklets created by the researchers based on Dietary Approaches to Stop Hypertension (DASH) diet as well as a self-management notebook we will provide to participants in which the they will record blood pressure, body weight and lifestyle improvement goals. The education booklets will be selected for that it will suitable for the individual participant. Any abnormalities in the monitored values or data or exacerbation of participant symptoms will be reported immediately to the primary care physician.

SMS content:

Diet Reduce sodium (salt) intake WHO recommended sodium intake is 5g/day Eat more fruits, vegetables and more fiber

Dietary Approaches to Stop Hypertension (DASH) eating plan:

It is high in fruits and vegetables, low-fat dairy, and fiber. Patients who strictly follow the DASH eating plan can also have fairly significant reductions in weight, particularly when combined with a low-sodium diet. Lifestyle, Stop smoking, Stop taking alcohol, Caffeine, Exercise: Regular exercise (walking, running) for 20 to 30 minutes most days of the week can lower your blood pressure, Reduce weight, Reduce stress, Monitor your blood pressure at home, Control blood pressure during pregnancy, Medication: Take medication regularly

Economic evaluation

Researchers have recommended with emphasis on economic evaluation of health promotion interventions such as health education and mobile health technology (SMS).

For this evaluation, the estimated cost of the program as well as costs for activities will be measured using ingredients approach, which includes listing of all types of inputs by identification of activities, quantities used, and prices for each input. Activity-based costing (ABC) techniques will be attempted to assign costs to each of the activities in the production process and/or resources. For this purpose, all costs will be classified according to major activities and/or resources. All activities and their associated inputs will be identified, and their respective costs will be obtained. Costs will be derived from two phases of the intervention named start-up cost and implementation cost which are directly related to the study. Total costs will be considered as the summation of capital and recurrent cost items for each phase. A comprehensive list of cost-related items will be made, and finally, cost per session per beneficiary will be estimated by dividing the total provider cost per session with the number of beneficiaries who received the SMS. The estimation of the cost will be covered the additional costs only that will include all field and administrative activities. Costs incurred other than intervention activities of the project such as salary, transportation, and data collection will be excluded from the estimation. Moreover, a household out of pocket expense/cost will be measured to assess any costs incurred for receiving the treatment or related to treatment. All necessary data will be extracted from the project's documents, and project staff members will be interviewed whenever necessary.

Objectives of the study are;

1. To capture the care seeking pattern due to chronic disease and other illness also.
2. To estimate the treatment cost from household perspectives due to chronic disease and other illness also.
3. To estimate the program cost from supply side perspective.
4. To conduct a Cost-Effectiveness Analysis (CEA) of the program.

Program costs/provider perspective

Start-up cost

Implementation cost

Household costs/household perspective

Cost-Effectiveness analysis

Cost-effectiveness ratio of the intervention package will finally be calculated using the cost of the whole program. Net cost of intervention and its effectiveness will be measured by comparing cost and effectiveness in intervention and control groups. Cost-outcome ratio as well as incremental cost-outcome ratio will be calculated i.e. if the study switches from one alternative (A) to another alternative (B), the changes in costs and outcomes will be compared (like, C1 - C0 / E1 - E0). Changes in various effects between intervention and comparison group will be considered as the changes in outcome/success of the intervention. The program with the low cost-effectiveness ratio will be considered as cost-effective intervention as it would offer most value for money.

Data management and analysis:

Data will be entered twice and stored in a relational database. Pre-coded questionnaire will be used to minimize data coding errors. All data forms and questionnaires will be checked for errors and necessary corrections will be made before data entry. A data entry program with built-in range and consistency checks will be used. Frequency distributions will be run to identify outliers. In all analyses, potential confounding variables and effect modifiers will be considered. Data will be entered, processed and analyzed using the statistical software packages SPSS for Windows version 21.0 and Epi Info version 7.0.

Statistical analyses will include descriptive as well as analytical methods. Basic presentations of data will include number and percentages of individuals with hypertension by age, sex and in relation to different known risk factors of interest. The descriptive statistics will be expressed as percentages, means, medians, standard deviations with ranges or with 95% confidence intervals where appropriate. Chi-square (χ2) tests will be computed to assess the association between outcome and independent variables. Odds ratios will be calculated for hypertension after adjusting for major confounding variables (e.g. age, sex, food habits, socioeconomic status, nutritional status, family history of hypertension etc.). Effects of interaction terms will also be examined fitting logistic regression models. When the main outcome measures are continuous variables, the statistical significance of group mean comparisons will be determined by Student's t-test. The primary analysis will be intention to treat which will provide relative unbiased comparisons among the intervention and control groups. In case of non-normal distribution of measurements, equivalent non-parametric tests will be used. Statistical significance will be defined as p<0.05. Secondary outcomes will be compared with the χ2 test for categorical outcome. Fisher's exact test when needed will be performed to estimate p values. For all models, the results will be expressed as an estimate of effect size, with 95% CIs and p values.

Outcome Variables:

Primary outcomes:

1. Behavioral changes by health education (evaluated by the researcher who developed questionnaire).

Operational Definition: Increased awareness, knowledge, and attitude changes will be measured by actual behavior change of participants. Once participants will aware the importance of lifestyle change, obtain knowledge about the way of change, and intend to change, the participants will change their lifestyles. Thus, we can measure these changes by actual behavior.

Secondary outcomes:

1. To decrease level of blood pressure
2. To measure health status by Euro-5D-5L QOL questionnaire (Mobility, self-care, usual activities, pain/discomfort, anxiety/depression)
3. To decrease dietary salt intake (Measured by food and urinary salinity test)
4. To measure blood glucose level (Random Blood Sugar), Urinary Protein and glucose test (In order to measure the complications)
5. Check the feasibility of mobile phone in hypertensive individuals by field testing questionnaires which will be developed by the researchers.

Ethical Implications:

The study will only be initiated after it has been approved by the Institutional Review Board (IRB) of Bangladesh Medical and Research Council (BMRC) as well as collaborating institutes in Bangladesh. Before enrolment, signed informed consent will be obtained from the participants. The consent form will be written in Bangla in a language and format that will be easily understood by the study participants of even little education. The consent form will be read out to the study participants. Signed consent or the left thumb impression will be obtained from the participants for participation in the study. A copy of the signed consent form will be given to the participant for their future questions and concerns. There will be some personal questions (age, income, contact address) for household respondents in the questionnaires. We will also collect blood and urine samples. So, there are some precautions will be taken to address the risk. Firstly, field researchers will be careful to emphasize the voluntary nature of engagement with the study and should ensure that participants will confirm written consent during the interview. Secondly, the personal questions will be asked in a calm and sensitive manner. Thirdly, during sample collection as much as possible we will take higher protection. Finally, total anonymity across all stages of the study will be maintained and access to raw data will be restricted to researchers only and stored securely.

ELIGIBILITY:
Inclusion Criteria:

1. Hypertensive individuals of either sex aged 35 years or older
2. Have 1-5 years of schooling
3. Resides within a radius of 3 miles from the Kumudini Women's Medical College and Hospital
4. Who resides in that area at least 6 months
5. Has a personal cell phone or access to a shared phone
6. Who is open and can exchange his views freely
7. Willing to participate in the study
8. Who consents to receive and read periodic text messages for the entire study period.

Exclusion Criteria:

1. Individuals with no hypertension aged less than 35 years
2. Who don't have 1-5 years of schooling
3. Resides beyond a radius of 3 miles from the Kumudini Women's Medical College and Hospital
4. Who don't reside in that area at least 6 months
5. With mental illnesses or serious co-morbidities or chronic illnesses that might cause periodic absence
6. Without access to cell phone
7. Not willing to participate
8. Who don't want to give consent to receive and read periodic text messages for the entire study period.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2018-08-12 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

PRIMARY OUTCOMES:
Behavioral change | Intervention period is 5 months
  By health education Operational Definition: Increased awareness, knowledge, and attitude changes will be measured by actual behavior change of participants. Once participants will aware the importance of lifestyle change, obtain knowledge about the way of change, and intend to change, the participants will change their lifestyles. Thus, we can measure these changes by actual behavior.
  Behavioral changes by health education (evaluated by the researcher who developed questionnaire).
  Operational Definition: Increased awareness, knowledge, and attitude changes will be measured by actual behavior change of participants. Once participants will aware the importance of lifestyle change, obtain knowledge about the way of change, and intend to change, the participants will change their lifestyles. Thus, we can measure these changes by actual behavior.
  Behavioral changes by health education (evaluated by the researcher who developed questionnaire).

SECONDARY OUTCOMES:
Improve quality of life | Intervention period is 5 months
  To decrease level of blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Jahan, Principal Investigator — Hiroshima University; Michiko Moriyama, Study Chair — Hiroshima University
Locations (1):
- Kumudini Women's Medical College and Hospital,, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jahan Y, Rahman MM, Faruque ASG, Chisti MJ, Kazawa K, Matsuyama R, Moriyama M. Awareness Development and Usage of Mobile Health Technology Among Individuals With Hypertension in a Rural Community of Bangladesh: Randomized Controlled Trial. J Med Internet Res. 2020 Dec 7;22(12):e19137. doi: 10.2196/19137. PMID 33284129
- [Derived] Jahan Y, Moriyama M, Rahman MM, Kazawa K, Rahman A, Sayeem Bin Shahid ASM, Das SK, Faruque A, Chisti MJ. Increasing Awareness and Use of Mobile Health Technology Among Individuals With Hypertension in a Rural Community of Bangladesh: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Aug 17;9(8):e15523. doi: 10.2196/15523. PMID 32804088